CLINICAL TRIAL: NCT07386145
Title: Whole-Body Vibration in Rehabilitation: Frequency and Voluntary Contraction-Dependent Activation of Tonic Vibration Reflex and Bone Myoregulation Reflex
Brief Title: Frequency and Voluntary Contraction-Dependent Activation of Tonic Vibration Reflex and Bone Myoregulation Reflex
Acronym: WBV-BMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nida dogan, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ND 2025-79
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Whole Body Vibration
Keywords: whole-body vibration; bone myoregulation reflex; tonic vibration reflex; muscle spindle; osteocyte; vibration; reflex latency

STUDY DESIGN:
Intervention Model Description: This is a crossover interventional study in which each participant is exposed to multiple whole-body vibration conditions with different frequencies and postures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-Frequency WBV - Upright Posture (Experimental): Participants will receive whole-body vibration at low frequencies (30, 32, 34, 36 Hz) while standing in an upright posture. Each vibration bout will last 15 seconds, with rest periods between trials. Soleus muscle activity will be recorded using surface electromyography during vibration.
  Interventions: Device: whole-body vibration
- Low-Frequency WBV - Semi-Squat Posture (Experimental): Participants will receive whole-body vibration at low frequencies while maintaining a semi-squat posture. Each vibration bout will last 15 seconds, with rest periods between trials. Soleus muscle activity will be recorded using surface electromyography during vibration.
  Interventions: Device: whole-body vibration
- High-Frequency WBV - Upright Posture (Experimental): Participants receive whole-body vibration at high frequency (40, 42, 44, 46 Hz) in an upright posture. Vibration will be applied in 15-second bouts with rest intervals.Soleus muscle activity will be recorded using surface electromyography during vibration.
  Interventions: Device: whole-body vibration
- High-Frequency WBV - Semi-Squat Posture (Experimental): Participants will receive whole-body vibration at high frequencies while standing in a semi-squat posture. Each vibration exposure will last 15 seconds, with rest intervals between trials. Soleus muscle activity will be recorded using surface electromyography during vibration.
  Interventions: Device: whole-body vibration

INTERVENTIONS:
Device: whole-body vibration — Participants will receive whole-body vibration using a vibration platform under different frequency and posture conditions. Vibration will be applied in short bouts (e.g., 15 seconds per trial) with rest periods between trials to minimize fatigue. Reflex and muscle activity responses will be recorded during vibration using surface electromyography (EMG)

SUMMARY:
When vibration is applied, sensors inside the muscle send signals to the nervous system, leading to automatic muscle activation. In this research, vibration will be applied using different body postures (such as standing or semi-squatting) and different vibration frequencies to understand how body position and vibration intensity influence muscle responses. Muscle activity will be recorded using surface electrodes placed on the skin. All procedures are non-invasive, painless, and do not involve medication or surgery.

The goal of this study is to improve understanding of how whole-body vibration affects muscle and nerve function. The findings may contribute to future rehabilitation strategies

DETAILED DESCRIPTION:
This study investigates how whole-body vibration (WBV) affects muscle reflex activity in healthy adults. Whole-body vibration will be delivered using a vibration platform that transmits mechanical oscillations through the lower limbs and trunk while participants maintain specific postures.

The primary objective is to examine how different vibration frequencies and different body postures influence reflex-related muscle activation. Secondary objectives include evaluating how vibration modifies neuromuscular excitability and the timing and magnitude of reflex responses.

Participants will be exposed to multiple experimental conditions across separate sessions. These conditions will include different postural tasks (such as upright standing and semi-squat) and different vibration frequencies, allowing comparison of how mechanical load distribution and sensory input alter reflex modulation. Each vibration application will last 15 seconds, and rest periods will be provided between trials to minimize fatigue and ensure measurement reliability.

Muscle activity will be recorded using surface electromyography (EMG) electrodes placed over the soleus muscle. Reflex responses under different postures and vibration frequencies will be recorded during vibration. Data processing and analysis will be performed offline after the experiment is completed.

This study is based on previous findings indicating that whole-body vibration can stimulate muscle spindle afferent receptors as well as osteocyte-related mechanoreceptors within bone tissue, thereby increasing afferent sensory input and transiently modulating spinal and supraspinal motor control mechanisms, including reflex excitability and motor unit recruitment patterns. By systematically varying posture and vibration frequency, the study aims to clarify how vibration-induced sensory input interacts with biomechanical and neural factors to shape reflex response behavior.

The findings obtained from this study are expected to contribute to a more effective and targeted use of whole-body vibration in neuromuscular training, balance rehabilitation, enhancement of movement performance, and support of bone health. Furthermore, the results are anticipated to provide a scientific basis for the development of optimized vibration-based intervention protocols that consider both neuromuscular and musculoskeletal effects in clinical and athletic settings.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-45 years old
* Volunteering to participate in the research

Exclusion Criteria:

* Refusal to participate in the study
* Intolerance to whole-body vibration (WBV)
* History of vertigo
* Presence of malignant disease
* Presence of chronic systemic disease
* Pregnancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-01-25 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Latency of the soleus reflex during whole-body vibration | Day 1 (During a single experimental session)
  The primary outcome measure is the latency of the soleus reflex activated by whole-body vibration (WBV). Reflex latency will be calculated using a cumulative averaging method. The vibration stimulus will be recorded via an accelerometer mounted on the vibration platform (LIS344ALH; ±6 g; ECOPACK®, Mansfield, TX, USA). The onset of the mechanical stimulus and the onset of the reflex response will be identified using cumulative averaging. Reflex latency will be defined as the time interval between the onset of the mechanical stimulus and the onset of the reflex response detected on surface electromyography (EMG), and will be expressed in milliseconds (ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Therapy and Rehabilitation Training Research Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided